CLINICAL TRIAL: NCT00565331
Title: A Prospective Randomized Study on the Efficacy and Safety of the Prophylactic Use of Rituximab, Added to Standard Immunosuppressive Treatment in Comparison With Standard Immunosuppressive Treatment Alone in Renal Transplantation
Brief Title: Rituximab for Prevention of Rejection After Renal Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry); Astellas Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRT06; UMC Radboud RI000131
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rituximab
  Interventions: Drug: Rituximab
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — single dose of rituximab of 375 mg/m2 intravenously at the time of transplantation
  Other Names: Mabthera, Rituxan
  Arms: 1
Drug: Placebo — saline solution
  Arms: 2

SUMMARY:
Our standard immunosuppressive treatment after renal transplantation is a combination of tacrolimus, mycophenolate mofetil, and prednisolone. With this regimen the incidence of acute rejection within the first six months after transplantation has dropped to about 20%. The main challenge at present remains to improve long-term outcome by preventing chronic allograft nephropathy (CAN). Since acute rejection is a strong predictor of CAN, a further decrease in the incidence of acute rejection can improve the long-term graft survival. Current strategies to prevent rejection are mainly directed at alloreactive T cells. Recently, the attention for the role of antibodies in the pathogenesis of acute rejection has increased. In addition, anti-B cell therapy was shown to be effective in diseases that were considered to be mainly T cell driven, like rheumatoid arthritis. In the latter case it has been suggested that anti-B cell antibodies may impair the antigen presenting function of B cells. We therefore decided to investigate the effectiveness and safety of the anti-B cell monoclonal antibody rituximab for prophylaxis of acute rejection after renal transplantation.

Study design: Double-blind, placebo controlled intervention study. One group receives a single dose of rituximab of 375 mg/m2 intravenously at the time of transplantation, and the other group receives a placebo infusion.

Primary Objective:

To determine the incidence and severity of biopsy-confirmed acute rejection within the first six months after transplantation.

Secondary Outcomes:

* Renal function as estimated by the endogenous creatinine clearance at 6 months
* Occurrence of chronic allograft nephropathy at 6 months
* Cumulative incidence of infections and malignancies at 6 months
* Medical costs during the first 6 months after transplantation
* Patient and graft survival

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients
* Signed, dated, and witnessed IRB approved informed consent

Exclusion Criteria:

* Pregnancy
* Living donor, who is HLA identical.
* Hemolytic uremic syndrome as original kidney disease.
* Focal segmental glomerulosclerosis that had recurred in a previous graft.
* More than two previously failed grafts and/or PRA > 85%.
* Previous treatment with anti-CD20 antibodies.
* Diabetes mellitus that is currently not treated with insulin.
* Total white blood cell count <3,000/mm3 or platelet count <75,000/mm3.
* Active infection with hepatitis B, hepatitis C, or HIV.
* History of tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of biopsy-confirmed acute rejection | First six months after transplantation

SECONDARY OUTCOMES:
Renal function as estimated by the endogenous creatinine clearance | 6 months after transplantation
Occurrence of chronic allograft nephropathy | First 6 months after transplantation
Cumulative incidence of infections and malignancies | First 6 months after transplantation
Patient and graft survival | First six months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Luuk Hilbrands, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Pescovitz MD. Rituximab, an anti-cd20 monoclonal antibody: history and mechanism of action. Am J Transplant. 2006 May;6(5 Pt 1):859-66. doi: 10.1111/j.1600-6143.2006.01288.x. PMID 16611321
- [Derived] Kamburova EG, Koenen HJ, van den Hoogen MW, Baas MC, Joosten I, Hilbrands LB. Longitudinal analysis of T and B cell phenotype and function in renal transplant recipients with or without rituximab induction therapy. PLoS One. 2014 Nov 13;9(11):e112658. doi: 10.1371/journal.pone.0112658. eCollection 2014. PMID 25393622
- [Derived] Smeekens SP, van den Hoogen MW, Kamburova EG, van de Veerdonk FL, Joosten I, Koenen HJ, Netea MG, Hilbrands LB, Joosten LA. The effects of in vivo B-cell depleting therapy on ex-vivo cytokine production. Transpl Immunol. 2013 Jun;28(4):183-8. doi: 10.1016/j.trim.2013.04.008. Epub 2013 May 4. PMID 23651756
- See also: Radboud University Nijmegen Medical Centre — http://www.umcn.nl/Pages/default.aspx